CLINICAL TRIAL: NCT05834790
Title: Effectiveness of Mobile Augmented Reality (MAR) on Oral Healthcare Education for the Independent Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MAR2023
Record Dates: First submitted 2023-03-13; First posted 2023-04-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-04

CONDITIONS: Aged

STUDY DESIGN:
Intervention Model Description: Three activity centers from the list will be randomly chosen and assigned to MAR, lecture, and no intervention groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MAR group (Experimental): The participants in this group will attend the MAR oral health education program
  Interventions: Other: Mobile Augmented Reality (MAR) for oral health education program
- lecture-based group (Active Comparator): The participants in this group will attend the lecture oral health education program
  Interventions: Other: Lecture-based oral health education program
- controlled group (No Intervention): The participants in this group will not attend any oral health education program

INTERVENTIONS:
Other: Mobile Augmented Reality (MAR) for oral health education program — MAR application named MAKAR will be available to download and use for smartphones and tablets. Participants will need to scan QR code to access the content of oral health education program
  Arms: MAR group
Other: Lecture-based oral health education program — The oral health education program that will be delivered by traditional lecture-based process
  Arms: lecture-based group

SUMMARY:
The goal of this clinical trial is to learn the outcomes of Mobile Augmented Reality (MAR) for oral health education program in the independent elderly. The main question it aims to answer is:

• Can MAR for oral health education program provide better outcomes comparing to lecture-based education program and no intervention group.

The activity centers from the list will be randomly chosen and assigned to MAR, lecture, and no intervention groups.

* Participants from activity centers that were assigned as MAR and lecture groups will attend one time education program. They have to finish questionnaires 3 times and receive 2 times oral examination.
* Participants from activity centers that was assigned as no intervention group will not attend any education program. They have to finish questionnaires 2 times and receive 2 times oral examination.

DETAILED DESCRIPTION:
Background/purpose: Aging is an inevitable global trend in this century. Elderly people are more susceptible to general health and oral health diseases which have negative impacts on their quality of life. Oral healthcare education could be the optimal measure to provide knowledge and develop self-care skills for elderly people to improve their oral health conditions. However, traditional passive lecture-based education programs might not be effective enough. There are many opportunities to improve the education program through digital technology. Mobile augmented reality (MAR) could be integrated into oral healthcare education to make education more effective. In this study, investigators would like to develop and evaluate the effectiveness of MAR-integrated oral healthcare education, as well as compare outcomes with traditional lecture-based education.

Materials and methods: Sixty independent elderly (age 65 or older) from six of Taipei city's local activity centers will be recruited. The participants will be required to be able to use smartphones in their daily life. The participants from one of the three activity centers will be randomly assigned to the MAR group (n=20), the other one activity centers will be assigned to the lecture group (n=20), and the rest will be assigned to the control group (n=20). The MAR group will be taught with MAR integrated education program, the lecture group will be taught with a traditional lecture-based program, while the control group will not undergo any education program. Outcome measurement will include oral healthcare knowledge, self-efficacy of oral healthcare, the usability of the MAR system, tongue coating, plaque index, and gingival index. The pre-, post-intervention, and two-weeks follow-up results will be compared by inferential statistics.

Results: The expected results are MAR integrated oral healthcare education could provide statistically significant improvement in participant outcomes compared to the control group and provide comparable or higher outcomes compared to the traditional education program. The usability score of MAR is acceptable.

Conclusion: MAR might be the feasible way to improve oral healthcare education for the independent elderly.

ELIGIBILITY:
Inclusion Criteria:

* the elderly who are able to use a smartphone
* the elderly who can read and understand traditional Chinese

Exclusion Criteria:

* the elderly who has communication problems

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Baseline oral healthcare-related knowledge | This outcome will be measured before intervention for all groups
  Fifteen statements will be used to measure participants' knowledge. The possible answers include True, False, and Don't know. Correct answer scores 1, while incorrect answer and Don't know score 0. A higher score indicates a higher degree of oral healthcare-related knowledge with a possible score of 0-15
Change of the baseline oral healthcare-related knowledge immediately after intervention | This outcome will be measured immediately after intervention for lecture and MAR groups
  Fifteen statements will be used to measure participants' knowledge. The possible answers include True, False, and Don't know. Correct answer scores 1, while incorrect answer and Don't know score 0. A higher score indicates a higher degree of oral healthcare-related knowledge with a possible score of 0-15
Change of the baseline oral healthcare-related knowledge 2 weeks after intervention | This outcome will be measured 2 weeks after intervention for all groups
  Fifteen statements will be used to measure participants' knowledge. The possible answers include True, False, and Don't know. Correct answer scores 1, while incorrect answer and Don't know score 0. A higher score indicates a higher degree of oral healthcare-related knowledge with a possible score of 0-15
Baseline self-efficacy about oral healthcare tools suitability evaluation and usage | This outcome will be measured before intervention for all groups
  Seven statements were used to evaluate participants' self-efficacy about oral healthcare tools' suitability evaluation and usage. Each item will be scored on a 5-point Likert-type scale ranging from 1, strongly disagree, to 5, strongly agree. A higher score indicates a higher degree of self-efficacy with a possible score of 7-35.
Change of the baseline self-efficacy about oral healthcare tools suitability evaluation and usage immediately after intervention | This outcome will be measured immediately after intervention for lecture and MAR groups
  Seven statements were used to evaluate participants' self-efficacy about oral healthcare tools' suitability evaluation and usage. Each item will be scored on a 5-point Likert-type scale ranging from 1, strongly disagree, to 5, strongly agree. A higher score indicates a higher degree of self-efficacy with a possible score of 7-35.
Change of the baseline self-efficacy about oral healthcare tools suitability evaluation and usage 2 weeks after intervention | This outcome will be measured before intervention for all groups
  Seven statements were used to evaluate participants' self-efficacy about oral healthcare tools' suitability evaluation and usage. Each item will be scored on a 5-point Likert-type scale ranging from 1, strongly disagree, to 5, strongly agree. A higher score indicates a higher degree of self-efficacy with a possible score of 7-35.

SECONDARY OUTCOMES:
Baseline tongue coating | This outcome will be measured before intervention
  Tongue coating will be determined by the Winkel tongue coating index (WTCI) which divides the tongue into 6 sections in total. The score in each section could be 0-2. A score of 0 means no tongue coating, a score of 1 means a light coating, and a score of 3 means heavy coating. The higher score will show the heavier coating on the participant's tongue, ranging from 0-12.
Change of the baseline tongue coating | This outcome will be measured 2 weeks after intervention
  Tongue coating will be determined by the Winkel tongue coating index (WTCI) which divides the tongue into 6 sections in total. The score in each section could be 0-2. A score of 0 means no tongue coating, a score of 1 means a light coating, and a score of 3 means heavy coating. The higher score will show the heavier coating on the participant's tongue, ranging from 0-12.
Baseline plaque index | This outcome will be measured before intervention
  The plaque index in this study will be recorded by using the modified plaque score (MPS). This system combined the O'Leary plaque control record and the Silness and Löe plaque index. The MPS will be evaluated at 4 sites (mesiobuccal, mid-buccal, distobuccal, and lingual) of 6 teeth (maxillary right first molar, maxillary right central incisor, maxillary left second molar, mandibular right second molar, mandibular left central incisor, and mandibular left first molar). A score in each site could be 0-3. A score of 0 means no plaque, a score of 1 means a film of plaque adhering to the free gingival margin and adjacent area of the tooth, a score of 2 means moderate accumulation of soft deposit, and a score of 4 means abundance of soft matter. The total score will be interpreted as an MPS percentage. The higher percentage will show the heavier plaque deposited.
Change of the baseline plaque index | This outcome will be measured 2 weeks after intervention
  The plaque index in this study will be recorded by using the modified plaque score (MPS). This system combined the O'Leary plaque control record and the Silness and Löe plaque index. The MPS will be evaluated at 4 sites (mesiobuccal, mid-buccal, distobuccal, and lingual) of 6 teeth (maxillary right first molar, maxillary right central incisor, maxillary left second molar, mandibular right second molar, mandibular left central incisor, and mandibular left first molar). A score in each site could be 0-3. A score of 0 means no plaque, a score of 1 means a film of plaque adhering to the free gingival margin and adjacent area of the tooth, a score of 2 means moderate accumulation of soft deposit, and a score of 4 means abundance of soft matter. The total score will be interpreted as an MPS percentage. The higher percentage will show the heavier plaque deposited.
Baseline gingival index | This outcome will be measured before intervention
  The Löe-Silness gingival index will be used to record the gingival status in this study. This system will be evaluated on 6 teeth (maxillary right first molar, maxillary right lateral incisor, maxillary left first bicuspid, mandibular right first molar, mandibular left lateral incisor, and mandibular right first bicuspid). A score in each tooth could be 0-3. A score of 0 means absence of inflammation, a score of 1 means mild inflammation, a score of 2 means moderate inflammation, and a score of 3 means severe inflammation. The average score will be calculated. The higher score will show more severe gingival inflammation, ranging from 0-3.
Change of the baseline gingival index | This outcome will be measured 2 weeks after intervention
  The Löe-Silness gingival index will be used to record the gingival status in this study. This system will be evaluated on 6 teeth (maxillary right first molar, maxillary right lateral incisor, maxillary left first bicuspid, mandibular right first molar, mandibular left lateral incisor, and mandibular right first bicuspid). A score in each tooth could be 0-3. A score of 0 means absence of inflammation, a score of 1 means mild inflammation, a score of 2 means moderate inflammation, and a score of 3 means severe inflammation. The average score will be calculated. The higher score will show more severe gingival inflammation, ranging from 0-3.

OTHER OUTCOMES:
Baseline Usability Scale | This outcome will be measured MAR group immediately after intervention
  The System Usability Scale (SUS) questionnaire is a commonly used questionnaire for evaluating usability.Ten statements were used with a 5-point Likert-type scale ranging from 1, strongly disagree, to 5, strongly agree. The scores will be assigned a rating using a curved grading scale (CGS).
Change of the baseline Usability Scale | This outcome will be measured MAR group 2 weeks after intervention
  The System Usability Scale (SUS) questionnaire is a commonly used questionnaire for evaluating usability.Ten statements were used with a 5-point Likert-type scale ranging from 1, strongly disagree, to 5, strongly agree. The scores will be assigned a rating using a curved grading scale (CGS).

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lun Hsu, Principal Investigator — National Yang Ming Chiao Tung University
Locations (6):
- Taiwan (6):
  - Guandu Elderly Activity Center, Taipei
  - Taoyuan Activity Center, Taipei
  - Datong Activity Center, Taipei
  - Hushan Village Activity Center, Taipei
  - Quanyuan village activity center, Taipei
  - Zhongxin Village Activity Center, Taipei

IPD SHARING:
Plan to Share IPD: No
investigators decided to not share IPD to other researchers